CLINICAL TRIAL: NCT00731523
Title: An Open-label, Single-dose, Parallel-group Study to Compare the Pharmacokinetics of FTY720 and Metabolites in Subjects With Severe Renal Impairment With That in Matched Healthy Control Subjects
Brief Title: Pharmacokinetics (PK) and Metabolism of FTY720 in Patients With Severe Renal Impairment and Healthy Matched Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFTY720D2108
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2011-02

CONDITIONS: Renal Insufficiency
Keywords: FTY720, Pharmacokinetics, Renal insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: fingolimod (FTY720)

INTERVENTIONS:
Drug: fingolimod (FTY720)

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of FTY720 and its metabolites in patients with severe renal insufficiency and in matched, healthy volunteers. This study will allow a better understanding of the effects of renal insufficiency on the disposition of FTY720.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subjects:

* Subjects must have a calculated glomerular filtration rate (GFR) by Cockcroft-Gault Equation ≥80 mL/min.

Severe Renal Impaired Patients:

* Patients not on dialysis with severe renal failure with a creatinine clearance < 30 mL/min as determined by Cockcroft-Gault Equation.
* Renal function should have been stable within the 3 months prior to study start.
* Patients with diabetes and/or hypertension who are in otherwise in good health may be included. However patients with diabetes must not have clinical evidence of gastropathy or enteropathy.

Exclusion Criteria:

All Subjects/Patients:

* History of multiple and recurring allergies or allergy to the investigational compound/compound class being used in this study
* History of retinal macular edema.
* History of any significant cardiovascular events such as myocardia infarction, valvular disease, angina, ischemic heart disease, dilated cardiomyopathy, dysrhythmia.
* History of immunocompromise, including a positive HIV (ELISA and Western blot) test result.

Severe Renal Impaired Patients:

* Use of any highly potent CYP3A4 inhibitor (e.g. erythromycin, ketoconazole, itraconazole) within 2 weeks prior to dosing.
* Use of beta blocker therapy within two (2) weeks prior to dosing.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
PK profile comparison between healthy volunteers and severe renal impaired patients, 3 weeks

SECONDARY OUTCOMES:
Assess the safety and tolerability, 3 weeks
Assess the influence of renal function on the pharmacokinetics of FTY720 metabolites M2 and M3, 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (1):
- Novartis Investigator Site, Moscow, Russia

REFERENCES:
- See also: Results for CFTY720D2108 can be found on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2749